CLINICAL TRIAL: NCT05040607
Title: Physical Fitness, Exercise Capacity and Activities of Daily Living in Primary Ciliary Dyskinesia: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hazal Sonbahar Ulu, MSc, PT, Hacettepe University
Other Study IDs: GO 19/730
Record Dates: First submitted 2021-08-24; First posted 2021-09-10 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-04

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome; Immotile Cilia Syndrome
Keywords: Primary Ciliary Dyskinesia; Kartagener Syndrome; Immotile Cilia Syndrome; Pulmonary Function; Respiratory Muscle Strength; Exercise Capacity; Physical Fitness; Inspiratory Muscle Strength Training
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Ciliary Dyskinesia (PCD): The first stage of the study:
  Data of 20 PCD patients from the database recorded between 10 July 2015 and 10 January 2017.
  The second stage of the study:
  -Data of 14 PCD patients who had lower inspiratory muscle strength from the same database underwent supervised inspiratory muscle training (IMT) with tapered flow resistive loading using Powerbreathe K5 device at our research unit and airway clearance techniques (ACT) as a home-based therapy for 6 weeks from the database recorded between 10 July 2015 and 10 January 2017.
  Interventions: Other: Data Collection
- Healthy Group: Data of 20 healthy subjects from the database recorded between 10 July 2015 and 10 January 2017.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — The first stage of the study:
  Retrospective data collection of pulmonary function, respiratory muscle strength, exercise capacity, physical fitness, and activities of daily living (ADL).
  The second stage of the study
  -Retrospective data of pulmonary function, respiratory muscle function, functional capacity before and after supervised inspiratory muscle training with POWERbreathe K5 device using tapered flow resistive loading and airway clearance techniques performed for 6 weeks in PCD with decreased respiratory muscle strength.
  Groups: Primary Ciliary Dyskinesia (PCD)
Other: Data Collection — -Retrospective data collection of pulmonary function, respiratory muscle function, exercise capacity, physical fitness, and activities of daily living (ADL).
  Groups: Healthy Group

SUMMARY:
Decreased pulmonary function, peripheral muscle strength, and exercise capacity were reported in primary ciliary dyskinesia (PCD) in recent studies. We aimed to investigate the data conducted between 10 July 2015 and 10 January 2015 of pulmonary function, respiratory muscle strength, exercise capacity, physical fitness, and activities of daily living (ADL) in PCD and healthy counterparts retrospectively at the first stage of the study and the effects of inspiratory muscle training on pulmonary function, respiratory muscle strength, and exercise capacity in PCD patients with decreased inspiratory muscle strength from the database recorded between 10 July 2015 and 10 January 2015 retrospectively at the second stage of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Being able to cooperate with the assessments
* Not having any orthopedic, or neurological problems

Exclusion Criteria:

* Not being clinically stable
* Not being able to cooperate with the assessments
* Having any orthopedic, or neurological problems

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient group: PCD patients consulted from Hacettepe University, Faculty of Medicine, Department of Pediatric Chest Diseases, Child Health and Diseases/, Ankara, Turkey to our unit for evaluation in terms of respiratory physiotherapy were included in our study.
  Healthy group: Healthy counterparts from our database of the previous studies were included in our study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
A primer outcome for the first stage of the study: Physical fitness | 10 July 2015-10 January 2015-retrospectively
  Munich Physical Fitness Test (MFT) was used to evaluate physical fitness. It is a test with six parameters including ball bounce, sandbag throwing, bending, vertical jumping, hanging and step test.
A primer outcome for the second stage of the study: Functional capacity | 10 July 2015-10 January 2015-retrospectively
  Functional capacity was evaluated with six minute walk test (6MWT).

SECONDARY OUTCOMES:
Demographic features | 10 July 2015-10 January 2015-retrospectively
  The age was recorded in years.
Demographic features | 10 July 2015-10 January 2015-retrospectively
  Weight was recorded in kilograms.
Demographic features | 10 July 2015-10 January 2015-retrospectively
  The length was saved in meters.
Demographic features | 10 July 2015-10 January 2015-retrospectively
  Body mass index was calculated by dividing the weight by the square of the height (kg/m^2) and recorded.
Pulmonary Function | 10 July 2015-10 January 2015-retrospectively
  Pulmonary function (FEV1 (forced expiratory volume in one second), FVC (forced vital capacity), FEV1/FVC, FEF25-75 (%) (forced expiratory volume 25-75 %) and PEF (peak expiratory flow)) assessed with a portable spirometer (Spirobank MIR, Italy).
Respiratory muscle functions | 10 July 2015-10 January 2015-retrospectively
  Respiratory muscle strength (maximal inspiratory pressure (MIP);maximal expiratory pressure (MEP), respectively) was measured with a portable, electronic mouth pressure monitor (Micro Medical MicroMPM, UK) and recorded.
  For second stage of the study; average inspiratory flow, inspiratory volume, and inspiratory work was evaluated based on the outcomes of the Breathe-Link software using POWERbreathe K5 device before and after IMT with tapered flow resistive loading and recorded.
Exercise Capacity | 10 July 2015-10 January 2015-retrospectively
  Exercise capacity was assessed with the modified shuttle walk test.
Activities of Daily Living | 10 July 2015-10 January 2015-retrospectively
  Glittre activities of daily living (ADL) test was used to evaluate daily life activity.

CONTACTS AND LOCATIONS:
Overall Officials: Hazal Sonbahar Ulu, MSc, Principal Investigator — Hacettepe University; Deniz Inal Ince, Prof. Dr., Study Chair — Hacettepe University; Deniz Inal Ince, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No